CLINICAL TRIAL: NCT04581603
Title: Cognitive Behavioral Therapy (CBT-I) Augmentation of Topiramate in Promoting Abstinence in Alcohol Use Disorder (AUD)
Brief Title: CBT-I Augmentation of Medication for Drinking in AUD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty recruiting patients
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Coatesville Veterans Affairs Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NURA-001-19F; I01CX001957 (NIH)
Record Dates: First submitted 2020-10-02; First posted 2020-10-09 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Use Disorder With Insomnia
Keywords: Alcoholism; Sleep Initiation and Maintenance Disorders; Cognitive Behavioral Therapy
MeSH Terms: conditions — Alcoholism; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Randomized, behavioral placebo-controlled trial.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: single-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MED + CBT-I (Active Comparator): This arm will consist of patients treated with topiramate, naltrexone, or topiramate + naltrexone on a clinical basis for 6 weeks and then randomized to Cognitive Behavioral Therapy for Insomnia (CBT-I). They will be continued on MED for the next 8 weeks of CBT-I treatment.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- MED + SHE (Placebo Comparator): This arm will consist of patients treated with topiramate, naltrexone, or topiramate + naltrexone for 6 weeks on a clinical basis for 6 weeks and then randomized to Sleep Hygiene Education (SHE). They will be continued on MED for the next 8 weeks of SHE treatment.
  Interventions: Behavioral: Sleep Hygiene Education

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — CBT-I is conducted weekly for eight sessions during which the subjects meet individual with the study clinician for 45 minutes on the first session and for 30 minutes for sessions 2-8. Session 1 serves as an orientation and the onset of Sleep Restriction Therapy. Sessions 2 & 3 deliver the three main components that include, Sleep Restriction Therapy, Stimulus control, and Sleep Hygiene. All the sessions excluding the last two sessions are dedicated to the titration of total sleep time and to ensure patient adherence. The fifth session is used to deliver a specific form of cognitive therapy. The final session is used to engage the patient in a relapse-prevention didactic (i.e., to review how insomnia becomes chronic and strategies that abort an extended episode of insomnia). The subject will return on week 9 to complete the post-intervention visit after 8 weeks of behavioral sleep treatment.
  Other Names: CBT-I
  Arms: MED + CBT-I
Behavioral: Sleep Hygiene Education — This non-active control arm of behavioral sleep intervention consists of psychoeducation on sleep hygiene, sleep-related disturbances, and the effects of stress on sleep that will be delivered weekly for 8 weeks, for a time duration that is identical to the CBT-I sessions. The effect of stress on sleep is a commonly used control condition in insomnia clinical trials. SHE is preferred to a monitor-only condition as it will control for contact with the therapist and elapsed time during sessions. The subject will return on week 9 to complete the post-intervention visit after 8 weeks of behavioral sleep treatment.
  Other Names: SHE
  Arms: MED + SHE

SUMMARY:
Alcohol Use Disorder (AUD) and insomnia are more prevalent in Veterans than in the general community. Furthermore, insomnia is comorbid in 36-91% of individuals with AUD and jeopardizes recovery by increasing their risk for relapse and complicating their clinical profile. The VA/DoD guidelines recommend four medications for the treatment of AUD by promoting abstinence and a reduction in drinking. Two of these medications (MED) used commonly are naltrexone and topiramate but they do not improve sleep continuity or insomnia. The recommended treatment for insomnia is Cognitive Behavioral Therapy for Insomnia (CBT-I), and it has shown efficacy in improving insomnia but with minimal benefit in improving abstinence. However, these studies have involved subjects in early or sustained remission. The proposed study will evaluate whether augmenting MED with CBT-I, after reducing drinking or achieving abstinence, bolsters recovery in AUD, by decreasing insomnia and improving abstinence. If this strategy shows good clinical results and the findings are replicated in a multi-center trial then the combination of MED with CBT-I should be considered a standard component of the initial management of AUD with insomnia.

DETAILED DESCRIPTION:
Alcohol Use Disorder (AUD) and insomnia are both more prevalent among Veterans than in the general population. While insomnia is 3-9 times more prevalent in AUD than in the general population, patients with comorbid AUD and insomnia suffer from higher severity of AUD with increased alcohol craving, reduced quality of life, impaired interpersonal functioning, higher risks for suicidal behavior and relapse during early abstinence. There are limited options to treat drinking behavior and insomnia due to side effect profile (disulfiram). Medications commonly used to treat pathological drinking and promote abstinence include Naltrexone and Topiramate. However, these medications do not improve insomnia. Furthermore, hypnotic medication treatments with trazodone, gabapentin, and ramelteon have shown variable impact for sleep disturbance and abstinence. By contrast, all four studies evaluating Cognitive Behavioral Therapy for Insomnia (CBT-I) have shown a large magnitude of effect for treating insomnia but with minimal to no effect on abstinence. Thus, combining MED and CBT-I will improve their insomnia and bolster their recovery. This combination treatment will be the first personalized intervention in treating Veterans with AUD and comorbid insomnia.

A sample of treatment-seeking Veterans with AUD (N=82) will be initially treated with a medication for drinking (MED), that will be either TOP 200 mg a day for six weeks, naltrexone 50 mg daily (and up to 100 mg daily), depot-naltrexone 380 mg injections every 4 weeks, or a combination of TOP + NTX. They will stabilized on the MED over 6 weeks and then randomized to receive either CBT-I (N=41) or Sleep Hygiene Education (SHE, a behavioral placebo intervention) (N=41) weekly for the next eight weeks. The investigators will conduct CBT-I following the standard protocol using 30-minute sessions to deliver its components (Sleep Restriction, Stimulus Control, Sleep Hygiene and Cognitive Therapy). A post-intervention visit will be conducted eight weeks after the end of the intervention phase. The primary outcome measure will be the the insomnia severity (as assessed using the Insomnia Severity Index). The secondary outcome measure will include the Percent Days Abstinent (as computed from the Time Line Follow Back interview). The investigators will also track other aspects of alcohol use, sleep and daily functioning using TLFB, PACS, sleep diaries, BDI, and the STAI to test whether successful treatment of drinking and insomnia will be associated with better clinical outcomes in AUD. It is hypothesized that in Veterans with AUD, the combination of MED+CBT-I, as compared to MED+SHE group, will lead to superior sleep-related outcomes along with pre-post treatment effect sizes comparable to the meta-analytic norms. On an exploratory basis, the MED + CBT-I arm will have a relatively higher percentage of days abstinent from alcohol and the improvement in insomnia and abstinence from drinking will show durability eight weeks after end of behavioral sleep treatment. If these hypotheses are supported, the findings will need to be validated in a larger multi-center trial. If validated, the findings would support: 1) including insomnia treatment as a standard component of the initial protocol for treating AUD comorbid with insomnia, and 2) using MED+CBT-I combination treatment to manage this subpopulation of AUD patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Veterans between the ages of 18 and 70 years.
* A past-year DSM-5 diagnosis of moderate to severe AUD (i.e., meeting 4 of the 11 DSM-5 criteria for AUD)
* Actively drinking alcohol within the past month ( 2 heavy drinking days, defined as 4 drinks/day for women and 5 drinks/day for men).
* Self-reported insomnia of moderate or severe intensity (i.e., an Insomnia Severity Index total score 15).
* Subject has expressed a desire to stop or reduce drinking.
* Capacity to comprehend and give informed consent.
* Women of child-bearing potential (i.e., who have not had a hysterectomy, bilateral oophorectomy, tubal ligation or is less than two years postmenopausal), must be non-lactating, practicing a reliable method of birth control, and have a negative urine pregnancy test prior to initiation of treatment.

Exclusion Criteria:

General

* A current, clinically significant physical disease or abnormality based on history, physical examination, or routine laboratory evaluation.
* Current serious psychiatric illness (i.e., schizophrenia, bipolar disorder, severe or psychotic major depression, eating disorder, or imminent suicide or violence risk).
* DSM-5 criteria for any other substance use disorder other than alcohol, nicotine, cannabis use disorder, or mild stimulant (cocaine) use disorder.
* Untreated subjects with a diagnosis of moderate-severe obstructive sleep apnea with a total Apnea Hypopnea Index (AHI-T) of 15 events/hour of sleep.
* Recent (within the 10 days prior to the baseline visit) exposure to licit or illicit opioids as defined by self-report or a positive urine drug screen. Individuals on a prescription low-dose opioid medication for chronic pain are eligible for treatment with TOP only, and positive urine drug screen(s) will not be exclusionary in this case.
* Patient also agrees not to initiate CBT for alcohol use disorder during the trial or will be discontinued.
* Completed a full course of CBT-I within the past year.

Specific to Naltrexone treatment

* A history of hypersensitivity to naltrexone.
* A transaminase elevation >300% of normal.
* Active treatment with opioid medications.

Specific to Topiramate treatment

* A history of hypersensitivity to TOP.
* A history of nephrolithiasis.
* A history of narrow angle glaucoma.
* Current treatment with medications considered a high risk for adverse reactions for TOP treatment, such as carbonic anhydrase inhibitors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index - Total Score | After eight weeks of behavioral sleep intervention
  Insomnia Severity Index (ISI): This 7-item (0-4 Likert scales) measure yields a total score of 28. The norms for the scale are as follows: 0-7 represents no clinically significant insomnia; 8-14 represents sub threshold insomnia; 15-21 represents clinical insomnia (moderate severity); 21-28 represents clinical insomnia (severe). The scale provides a measure of severity of insomnia (overall), a measure of insomnia subtype, a measure of the diurnal effects of insomnia, and a measure of sleep "satisfaction". The ISI will be completed at baseline and for all the subsequent study-related visits.

SECONDARY OUTCOMES:
Change in Percent Days Abstinent (PDA) on the Time Line Follow Back Measure | After eight weeks of behavioral sleep treatment
  Time Line Follow Back measure (TLFB): The TLFB provides assessment of drinking using a calendar format for the number of standard alcoholic beverages consumed per day. A standard drink, as defined by the National Institutes of Health, is 12 oz of regular beer, 5 oz of regular wine, or 1.5 oz of distilled spirits (e.g. whiskey). Numerous indices may be derived from the TLFB, such as the Percent Days Abstinent (PDA) proposed in this study. The PDA is derived as the percentage of days an individual reports being abstinent from alcohol within a given assessment time period.
Change in Percent Days Abstinent (PDA) on the Time Line Follow Back Measure | Eight weeks after end of behavioral sleep intervention (about 17 weeks since start of behavioral sleep treatment)
  Time Line Follow Back measure (TLFB): The TLFB provides assessment of drinking using a calendar format for the number of standard alcoholic beverages consumed per day. A standard drink, as defined by the National Institutes of Health, is 12 oz of regular beer, 5 oz of regular wine, or 1.5 oz of distilled spirits (e.g. whiskey). Numerous indices may be derived from the TLFB, such as the Percent Days Abstinent (PDA) proposed in this study. The PDA is derived as the percentage of days an individual reports being abstinent from alcohol within a given assessment time period.
Change in Insomnia Severity Index - Total Score | Eight weeks after end of behavioral sleep intervention (about 17 weeks since start of behavioral sleep treatment)
  Insomnia Severity Index (ISI): This 7-item (0-4 Likert scales) measure yields a total score of 28. The norms for the scale are as follows: 0-7 represents no clinically significant insomnia; 8-14 represents sub threshold insomnia; 15-21 represents clinical insomnia (moderate severity); 21-28 represents clinical insomnia (severe). The scale provides a measure of severity of insomnia (overall), a measure of insomnia subtype, a measure of the diurnal effects of insomnia, and a measure of sleep "satisfaction". The ISI will be completed at baseline and for all the subsequent study-related visits.

CONTACTS AND LOCATIONS:
Overall Officials: Subhajit Chakravorty, MD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (2):
- United States (2):
  - Coatesville VA Medical Center, Coatesville, PA, Coatesville, Pennsylvania
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT04581603/ICF_000.pdf